CLINICAL TRIAL: NCT03114670
Title: Donor-derived Anti-CD123 Chimeric Antigen Receptors Modified T Cells for Recurred Acute Myeloid Leukaemia After Allogeneic Hematopoietic Stem Cell Transplantation
Brief Title: Donor-derived Anti-CD123-CART Cells for Recurred AML After Allo-HSCT
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Affiliated Hospital to Academy of Military Medical Sciences (Other)
Responsible Party: Principal Investigator, Chen Hu, Affiliated Hospital to Academy of Military Medical Sciences, Affiliated Hospital to Academy of Military Medical Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 307-RV-CAR-123
Record Dates: First submitted 2017-03-21; First posted 2017-04-14 (Actual); Last update posted 2017-06-14 (Actual); Status verified 2017-06

CONDITIONS: Adult Acute Myeloid Leukemia
Keywords: Leukemia; Leukemia, Myeloid; Recurrence; Neoplasms by Histologic Type; Disease Attributes; Cyclophosphamide; Fludarabine; CD123; Chimeric Antigen Receptor modified T-cells
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Leukemia; Leukemia, Myeloid; Recurrence; Neoplasms by Histologic Type; Disease Attributes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- CD123CAR-41BB-CD3zeta-EGFRt-expressing T cells (Experimental): Patients will receive a full dose CART infusion at day 0.
  Interventions: Biological: CD123CAR-41BB-CD3zeta-EGFRt-expressing T cells

INTERVENTIONS:
Biological: CD123CAR-41BB-CD3zeta-EGFRt-expressing T cells — a single dose of CD123CAR-41BB-CD3zeta-EGFRt-expressing T cells will be infusion after preconditioning.
  Other Names: anti-CD123 CART, CART123

SUMMARY:
Patients with acute myeloid leukemia(AML) recurred after the allogeneic hematopoietic stem cell transplantation (allo-HSCT) have a dismal prognosis.The investigators developed donor-derived chimeric antigen receptor modified-T cell(CART) to target CD123 for the treatment of AML. The investigators start the Phase I study aimed to treat recurred post-transplantation AML patients using donor-derived CAR-T. The purpose of this study is to assess the safety and effectiveness of anti-CD123 CAR-T cells in patients.

DETAILED DESCRIPTION:
Allo-HSCT is increasingly being used for AML, however, leukemia relapse remain a main problem for decades.Recently the investigators have witnessed great progresses in cancer therapy with chimeric antigen receptors modified T cells(CAR-T), especially for B-cell malignance. preclinical data about anti-CD123 CART have shown raised serious safety concerns of human anti-CD123 CAR-T for severe impairment of normal hematopoiesis in NSG mice.Patients with AML recurred after allo-HSCT have a dismal prognosis.The investigators developed donor-derived CART to target CD123 for the treatment of AML. The investigators start the Phase I study aimed to recurred post-transplantation AML patients using donor-derived CAR-T. The purpose of this study is to assess the safety and effectiveness of anti-CD123 CAR-T cells in patients.

ELIGIBILITY:
Inclusion Criteria:

1. Male and Female subjects with CD123+ acute myeloid leukemia as confirmed by immunohistochemistry and flow cytometry;
2. Patients must have received an allogenic stem cell transplantation(Allo-HSCT). The leukemia relapsed. There are available donor or enough cryopreserved donor-derived PBMCs for CART preparation and subsequent Allo-HSCT. In the previous case, the donor should have adequate venous access for apheresis.
3. Karnofsky score greater than 70%;
4. patients more than 18 years of age
5. Expected survival time >16 weeks;
6. Bilirubin <3.0 mg/dL,
7. Alanine aminotransferase(ALT)/ aspartate aminotransferase(AST)<3 fold normal.
8. Diffusing capacity of the lung for carbon monoxide(DLCO) and forced expiratory volume in one second(FEV1)>45% of predictive value.
9. At least received three kinds of medicines functioning by different mechanisms, including alkylating agents, protease inhibitors, and immunomodulators, and disease progressing within 60 days.
10. Important organs are well tolerated;
11. For post-transplantation patients, the apheresis would be undertaken only at least 2 weeks after immunosuppressive agents for GvHD withdrawal;
12. From very beginning of the test to 30 days after the withdrawal, men and women should adopt reliable contraceptive measures.
13. All research participants must have the ability to understand and willingness to sign a written informed consent.

Exclusion criteria:

1. Patients were diagnosed with APL M3:t(15; 17)(q22; q12);PML/RARα ）；
2. Symptomatic active central nervous system leukaemia;
3. Patients with HIV, hepatitis B or C infection;
4. Any concurrent active malignancies;
5. Other uncontrolled active illness that hinders participation in the trial;
6. Patients suffer from coronary heart disease, angina pectoris, myocardial infarction, arrhythmia, cerebral thrombosis, cerebral hemorrhage and other serious heart, cerebrovascular disease;
7. patients with poorly controlled hypertensive
8. patients with froward psychiatric history
9. anyone who the researchers think unsuitable to participate in the investigation;
10. anyone who long-term use of immunosuppressive agents for organ transplants or other reasons, or undertake inhaled corticosteroids therapy recently.
11. failed production release testing: CAR+ T cells <30% or T cell expansion less than 5-fold under the CD3/28 beads stimulation.
12. Pregnant, lactating or female patients planning to get pregnant within 2 months before treatment ends;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-03-25 (Actual); Primary Completion 2019-03-18 (Estimated); Study Completion 2021-03-18 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events related to treatment as assessed by NCI CTCAE version 4.03 | 15 years

SECONDARY OUTCOMES:
CART cells persistence in vivo | 15 years
CAR123-specific antibody level | 15 years
Overall survival | 15 years
Disease response(CR, CRi) | 15 years

CONTACTS AND LOCATIONS:
Overall Officials: Hu Chen, M.D., Ph.D., Study Director — Affiliated Hospital to Academy of Military Medical Sciences, China
Locations (1):
- Fengtai District, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided